CLINICAL TRIAL: NCT02355392
Title: Prevalence of Hypertension Using Telemedical Home Blood Pressure Measurements
Status: Completed | Type: Observational
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, Professor, Chief Physician, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Other Study IDs: M-20110011
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Telemedical home blood pressure measurements

SUMMARY:
The purpose of this study is to determine the prevalence of hypertension among citizens of Holstebro, Denmark aged 55-64 years, including both the well treated, the untreated and the insufficiently treated, and to estimate the prevalence of white coat and masked hypertension using home blood pressure measurements with telemedical data transmission.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 to 64 years
* Registered address in the municipality of Holstebro
* Enrolment at a practice of one of the GPs who had agreed to participate in the study.

Exclusion Criteria:

* Unwillingness to participate
* Incapability to do home blood pressure measurements

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A population study in the municipality of Holstebro, which has 57.000 inhabitants. Using the Civil Registration System, we invite all citizens aged 55-64 years.
Sampling Method: Non-Probability Sample
Enrollment: 3159 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Office blood pressure | 10 minuttes
Telemedical home blood pressure | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai Hoffmann-Petersen, MD, Principal Investigator — Department of Medical Research and Medicine, Holstebro Regional Hospital, Holstebro, Denmark

REFERENCES:
- [Derived] Hoffmann-Petersen N, Lauritzen T, Bech JN, Pedersen EB. High Prevalence of Hypertension in a Danish Population Telemedical Home Measurement of Blood Pressure in Citizens Aged 55-64 Years in Holstebro County. Am J Hypertens. 2016 Apr;29(4):439-47. doi: 10.1093/ajh/hpv116. Epub 2015 Jul 23. PMID 26208671